CLINICAL TRIAL: NCT00238459
Title: Immunopathogenesis of Acute and Early HIV Infection and the Role of HIV-Specific CD4 T Cell Responses and the Effect of Their Enhancement by Potent Antiretroviral Drugs and an HIV Vaccine Adequate Vaccine Was Not Provided.
Brief Title: Controlling Acute or Early HIV Infection With Antiretroviral Drugs, Without a Candidate Vaccine.As Reported Previously, the Candidate Vaccie Was Not Provided by the Maufacturer as Promised
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Fred T. Valentine, Professor of Medicine, National Institute of Allergy and Infectious Diseases (NIAID)
Other Study IDs: 5P01AI57127-2; 5P01AI057127 (NIH)
Record Dates: First submitted 2005-10-11; First posted 2005-10-13 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: HIV Infections
Keywords: Immunity to HIV; Acute Infection; Treatment Naive; Treatment Interruption; Structured Treatment Interruption; STI
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sequential samples from patients with acute and recent HIV infection
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Recently infected patients: Cohort 1)Patients elcted to be immediately treated with licensed drugs:21 patients Cohort 2) Or to delay treatment until clinically indicated:16 patieints
  Interventions: Drug: multiple licensed drugs not randomized
- A vaccine,HIV-1 immunogen was not provided for evaluation: In the intial design, acandiate HIV vaccine was to be evaluated, but in August 2007 the manufacturer refused to provide vaccine to allow this study to evaluate the effect of a vaccine on control of HIV. Therefore the study became an observational study of the effects of early versus delayed initiation of antiretrovral therapy on the preservation of anti-HIV immune responses and the ability of patients to control virus after a closely monitored discontinuation of therapy.
  Interventions: Drug: Patients elected to take licensed drugs. The vaccine was not provided for evaluation; Drug: multiple licensed antiretroviral drugs; not randomized; Other: Intended vaccine not provided, Licensed drugs provided, but were not investigated

INTERVENTIONS:
Drug: Patients elected to take licensed drugs. The vaccine was not provided for evaluation — Note:In August 2007 we were notified by the manufacturer that the experimental vaccine was no longer being made and would no longer be available for this study. Too few participants have received the vaccine or placebo to conclude anything about potential efficacy
  Groups: A vaccine,HIV-1 immunogen was not provided for evaluation
Drug: multiple licensed drugs not randomized
  Groups: Recently infected patients
Drug: multiple licensed antiretroviral drugs; not randomized
  Groups: A vaccine,HIV-1 immunogen was not provided for evaluation
Other: Intended vaccine not provided, Licensed drugs provided, but were not investigated
  Groups: A vaccine,HIV-1 immunogen was not provided for evaluation

SUMMARY:
The purpose of this study is to determine the role of HIV-specific CD4 T cell responses and immune responses dependent upon these CD4 responses that develop when antiretroviral drugs are started during acute or recent HIV infection, whether these CD4 responses can be enhanced with a therapeutic HIV vaccine (HIV-1 immunogen), and what pattern of HIV-specific immune responses is associated with control of HIV upon discontinuation of antiretroviral drugs during an analytical therapeutic interruption. Participants will be treatment-naive adults with acute or early HIV infection who will choose to start or not start anti-HIV drugs at the beginning of the study. NOTE: In August 2007 we were notified by the manufacturer of the candidate vaccine that they were no longer making the vaccine, and that the vaccine would no longer be available. Unfortunately too few participants have received either the vaccine or placebo to conclude anything about efficacy. No safety problems occurred.

DETAILED DESCRIPTION:
In some HIV patients with acute or early infection, effective long-term immunological control of HIV occurs, indicating that before HIV caused irreparable damage, their immune systems were able to mount an effective immune response to HIV. However, it is unknown how the immune systems of such patients with acute or early infection are able to develop and maintain effective memory CD4 immune responses. In other HIV patients, it is the destruction of CD4 cells and an ever-weakening immune system that leads to the progression of HIV disease. HIV-1 immunogen is a whole killed gp120-depleted HIV vaccine composed of an HIV-1 isolate (HZ321) from serum collected from a patient in Zaire in 1976. The vaccine contains proteins from HIV subtypes A and G. By injecting these particles into HIV infected people, the immune system may be stimulated to mount a greater immune response not only to the killed HIV particles of the vaccine but also to real virus particles and HIV infected cells in these people. Also, because HIV-1 immunogen is based on whole inactivated virus, it may stimulate broader immune responses that are capable of suppressing more diverse HIV strains than currently available vaccine preparations that are based on single subunit proteins of HIV. This study was planned to evaluate the safety and efficacy of a therapeutic HIV vaccine, HIV-1 immunogen, in conjunction with STIs, in controlling HIV infection during acute or early infection. Participants will be antiretroviral therapy (ART)-naive and will choose to either start or not start ART in this study.

Participants will elect to start or not start ART at the start of this study. Those participants who choose not to begin ART will not receive any intervention during this study but will be followed for the entire length of the study. Those participants that choose to begin ART will start taking study-approved ART in Step 1 of the study. Only patients who have a viral load of less than 50 copies/ml by Week 24 will proceed to Step 2; all other patients who begin ART will continue on study-approved ART but will not receive any vaccinations over the course of the study. Step 2 is the STI part of the study. In Step 2, patients will stop ART and will be randomly assigned to receive therapeutic vaccine or placebo injections at three timepoints: at the start of Step 2 and 12 and 24 weeks after starting Step 2. Injections will be given only to patients who have been on ART for at least 48 weeks; patients will receive their assigned injections 36 weeks after their first viral load reading of less than 50 copies/ml. A patient will enter Step 3 after having restarted ART for a minimum of 8 weeks after Step 2 ends, when the patient's viral load is less than 400 copies/ml and CD4 count is greater than 250 cells/ml. Entry into Step 4, which will include additional retreatment and revaccination, may be necessary for some participants, depending on individual immune response to the study-given ART and the injections.

The ART participants in this study will receive either study-provided ART or another approved ART; however, only study-provided ART will be provided by the study. Viral load and CD4 count will be closely monitored and will guide retreatment and revaccination as necessary. Blood collection will occur at all visits. A physical exam will occur at most visits. Urine collection and quality of life and adherence questionnaires will occur at selected visits.

NOTE: In August 2007 we were notified by the manufacturer of the candidate vaccine that they were no longer making the vaccine, and that the vaccine would no longer be available. Unfortunately too few participants have received either the vaccine or placebo to conclude anything about efficacy. No safety problems occurred.

ELIGIBILITY:
Inclusion Criteria:

* Acute or early HIV infection
* ART naive
* Willing to use acceptable forms of contraception

Exclusion Criteria:

* Allergy/sensitivity to any components of the vaccine
* Currently involuntarily incarcerated
* Pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acutely HIV infected patients: virus positive antibody negative Recently HIV infected patients: virus positive, low titers of antibody
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2005-07; Primary Completion 2011-03 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Effects of treatment on HIV-specific immune responses. | Weekly and then monthly after stopping antiretroviral drugs

SECONDARY OUTCOMES:
Immune control of HIV after stopping antiretroviral drugs. | Weekly and then monthly after stopping antirretroviral drugs

CONTACTS AND LOCATIONS:
Overall Officials: Fred Valentine, MD, Principal Investigator — NYU Langone Health
Locations (2):
- New York University School of Medicine, New York, New York, United States
- McGill University and University of Montreal, Montreal, Quebec, Canada

REFERENCES:
- [Background] Peters BS. The basis for HIV immunotherapeutic vaccines. Vaccine. 2001 Dec 12;20(5-6):688-705. doi: 10.1016/s0264-410x(01)00394-2. PMID 11738732
- [Background] Stekler J, Collier AC. Primary HIV Infection. Curr HIV/AIDS Rep. 2004 Jun;1(2):68-73. doi: 10.1007/s11904-004-0010-2. PMID 16091225
- [Background] Wahren B, Liu M. Therapeutic vaccination against HIV. Expert Rev Vaccines. 2004 Aug;3(4 Suppl):S179-88. doi: 10.1586/14760584.3.4.s179. PMID 15285716
- See also: Click here for more information about the Center of AIDS Research at the New York University School of Medicine — http://www.HIVinfosource.org